CLINICAL TRIAL: NCT06017752
Title: Development, Acceptability, and Short-Term Outcomes of a Teacher Module for a Brief, Bullying Bystander Intervention for Middle School Students in Rural, Low-Income Communities
Brief Title: Middle School Teacher Module for a Brief Bullying Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: Mental Research Institute (Other)
Responsible Party: Principal Investigator, Aida Midgett, Professor, Boise State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101-SB20-174
Record Dates: First submitted 2023-08-22; First posted 2023-08-30 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Bullying
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAC Teacher Module (Experimental)
  Interventions: Behavioral: STAC Teacher Module

INTERVENTIONS:
Behavioral: STAC Teacher Module — The STAC Teacher Module is a 30-minute presentation that includes normative feedback, didactic information, a review of the student STAC strategies and corresponding strategies teachers can use to support students who act as defenders, and information about "perceptions vs. facts" about bullying.

SUMMARY:
This study evaluates the feasibility and short-term outcomes of a teacher training designed as a companion module to a bullying bystander intervention (STAC) for middle school students in rural communities. The aim of this project is to provide a brief, low-cost intervention that can be easily disseminated as part of a school-based bullying prevention program to address this important public health problem.

ELIGIBILITY:
Inclusion Criteria:

* Being a teacher of an adolescent enrolled in grades 6, 7, or 8 in a participating middle school in Idaho.
* Speaks and reads English.
* Consents to participate.

Exclusion Criteria:

* Speaks and reads only a language other than English.
* Does not consent for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boise State Univerity, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STAC Teacher Module
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.76 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Knowledge and Confidence to Support Defenders
Description: Teacher-Advocates Pre- and Post-Scale (TAPPS) Knowledge and confidence to support defenders was measured using the TAPPS. The TAPPS is an 11 item survey that measures knowledge of buying behaviors, knowledge of how to support students using the STAC strategies, and confidence supporting students who intervene in bullying situations. Items are rated on a 4-point Likert Scale ranging from 1 (Totally Disagree) to 4 (Totally Agree) and were summed to compute a total scale score.
  Minimum =11; Maximum = 44 Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (50 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
score on a scale
  Pre-Test | 30.71 (2.95)
  Post-Test | 37.34 (3.90)

2. Primary Outcome: Confidence Managing Bullying
Description: Teacher's Attitudes about Bullying Questionnaire Confidence about managing bullying was measured using the Teacher's Attitudes about Bullying Questionnaire. This questionnaire is a 22 item survey. The 3-item Confidence in Managing Bullying Subscale was used. Items are rated on a 5-point Likert Scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) and are summed to compute a total scale score.
  Minimum = 3; Maximum = 15 Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (50 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
score on a scale
  Pre-Test | 10.47 (1.70)
  Post-Test | 13.12 (1.54)

3. Primary Outcome: Comfort Managing Bullying
Description: National Education Association Bullying Survey Comfort with managing bullying was measured using items from the National Education Association Bullying Survey. Participants were asked "How comfortable would the participant feel intervening when the participant sees the following bullying behaviors?" followed by five types of bullying (a) Physical, (b) Verbal, (c) Relational, (d) Cyberbullying , and (e) Sexting. Items are rated on a 5-point Likert Scale ranging from 1 (Very Uncomfortable) to 5 (Very Comfortable) and are summed to compute a total scale score.
  Minimum = 5; Maximum = 25 Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (50 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
score on a scale
  Pre-Test | 11.42 (1.62)
  Post-Test | 13.06 (1.95)

4. Primary Outcome: Bullying Self-Efficacy
Description: Bullying Self-Efficacy Teachers' self-efficacy in handling bullying situations was measured by two items from the National Education Association Bullying Survey. The items are rated on a 4-point Likert Scale ranging from 1 (Strongly Disagree) to 4 (Strongly Agree) and are summed to compute a total scale score.
  Minimum = 2; Maximum = 8 Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (50 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
score on a scale
  Pre-Test | 4.65 (0.86)
  Post-Test | 6.82 (1.01)

5. Primary Outcome: Number of Participants Reporting a Score of 4 or 5 on Intention to Use Teacher STAC Strategies
Description: The intention to use Teacher STAC strategies was measured using an adapted version of the Use of STAC Strategies for students. Items were adapted from the student version to be appropriate for teachers. The 4-item measures asks teachers "How likely the participant is to support students using these strategies to intervene in bullying in the future?: a) Stealing the Show - support students using humor or distraction to get the attention away from the bullying situation, b) Turning it Over - support a student who reported bullying to the participant or supporting students to report to a principal or School Resource Officer (SRO), c) Accompanying Others - support students who reach out to the student who was the target of bullying, or d) Coaching Compassion - support students who help the student who bullied develop empathy for the target." Items are rated on a 5-point Likert Scale ranging from 1 (Very Unlikely) to 5 (Very Likely).
Time Frame: immediate post-training (50 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
Participants
  Stealing the Show | 16
  Turning it Over | 16
  Accompanying Others | 17
  Coaching Compassion | 14

6. Secondary Outcome: Number of Participants Reporting a Score of 3 or 4 on Acceptability and Relevance of the Teacher STAC Training
Description: Program acceptability (e.g., how easy the program is to understand, utility of the program, program characteristics including interesting content and relevance of information presented, participant learning, and interest in recommending program to others) was assessed using a social validity survey composed of 8 items. Items were ranked on a 4-point scale from 1 (Strongly Disagree) to 4 (Strongly Agree).
Time Frame: immediate post-training (50 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Teacher Module
Number analyzed (Participants) | 17
Participants
  Easy to understand | 16
  Useful | 16
  Interesting | 15
  Relevant information | 15
  Relevant examples | 16
  Relevant role-plays | 16
  Learned something | 16
  Would recommend | 16

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | STAC Teacher Module
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT06017752/Prot_SAP_000.pdf